CLINICAL TRIAL: NCT04961593
Title: Pharmacokinetics and Pharmacodynamics of Caspofungin in Children Severe Infection
Brief Title: PK/PD of Caspofungin in Children Severe Infection
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-24
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pharmacokinetics; Infection, Fungal
MeSH Terms: conditions — Mycoses | interventions — Caspofungin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: Children treated with caspofungin in the pediatric intensive care unit
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — For children 3 months of age, the recommended dose is 70 mg/m2 for load and then 50 mg/m2 for maintenance, intravenous injection, once daily up to 5 days.

SUMMARY:
Caspofungin is an anti-fungal drug mainly metabolized by the liver. The pathophysiological status of children with severe infection will affect the metabolism of caspofungin in the body especially in the case of liver dysfunction. There is little metabolism of caspofungin through the kidney and continuous renal replacement therapy and renal function have little influence on the pharmacokinetics of caspofungin. The study aim to investigate PK/PD of caspofungin in children with specific pathophysiological conditions, such as liver insufficiency, hypoproteinemia, ECMO treatment, or sepsis.

DETAILED DESCRIPTION:
The current international recommended dose of caspofungin is 70 mg per square metre for load for children who is older than three months of age, followed by 50 mg per square metre for maintenance. For newborns and infants younger than 3 months of age，25 mg per square metre is also recommended.

Whether such a recommended dose can achieve an ideal PK/PD target in children with liver insufficiency, hypoproteinemia, ECMO treatment, or severe infection is still lacking in sufficient clinical data.

The objective of this study is to investigate PK/PD of caspofungin in children with specific pathophysiological conditions, such as liver insufficiency, hypoproteinemia, ECMO treatment, or sepsis.

Blood sampling time points of caspofungin are listed as follow:

Before administration (0 min); 1 h, 2 h, 4 h, 8 h , 12 h and 24 h after administration.

The concentration of caspofungin in whole blood will be analyzed at Huashan Hospital of Fudan University.

ELIGIBILITY:
Inclusion Criteria:

* Children receiving caspofungin in pediatric intensive care unit

Exclusion Criteria:

* No Informed Consent signed Participate in other clinical trials

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children receiving caspofungin in pediatric intensive care unit including but not limited to children with liver insufficiency, hypoproteinemia, ECMO treatment, CRRT treatment or sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) Pharmacokinetic Parameter | Day 1-5
  Time to reach the maximum plasma concentration (Tmax) after administrations of a single dose and multiple doses of the study drug

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration Pharmacokinetic Parameter | Day 1-5
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration after administrations of a single dose and multiple doses of the study drug
AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity Pharmacokinetic Parameter | Day1-5
  Area under the plasma concentration-time curve from time 0 to infinity after administration of a single dose of the study drug.
AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Pharmacokinetic Parameter | Day1-5
  Area under the curve from 0 to 24 hours after administrations of a single dose and multiple doses of the study drug.
Terminal Phase Elimination Half-life (T1/2) Pharmacokinetic Parameter | Day1-5
  Time required for half of the drug to be eliminated from the plasma after administration of a single dose of the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Lu, doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu N, Shi Y, Ju G, Liu X, Yan G, Zheng Y, Hou S, Xiang X, Lu G, Ouyang D, Zhu X, Wang Y. Population pharmacokinetics of caspofungin in critically ill Chinese children: a prospective observational study. Antimicrob Agents Chemother. 2025 Dec 30:e0127725. doi: 10.1128/aac.01277-25. Online ahead of print. PMID 41468548